CLINICAL TRIAL: NCT02259023
Title: Discretionary Food Sources and Stress Perception
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: DFS2014
Record Dates: First submitted 2014-09-29; First posted 2014-10-08 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Stress Perception; Discretionary Calories; Over All Health
Keywords: Stress Perception; Discretionary Calories; Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Liquid: Sugar sweetened beverage consumption (Experimental): Consumption of sugar-sweetened beverages
  Interventions: Other: Liquid: Sugar sweetened beverage consumption; Other: Solid: Grain based desserts and candy consumption
- Solid: Grain based desserts and candy consumption (Experimental): Consumption of grain based desserts and/or candy
  Interventions: Other: Liquid: Sugar sweetened beverage consumption; Other: Solid: Grain based desserts and candy consumption

INTERVENTIONS:
Other: Liquid: Sugar sweetened beverage consumption — Sugar sweetened beverage consumption
Other: Solid: Grain based desserts and candy consumption — Grain based desserts and candy consumption

SUMMARY:
Purpose:

The objective of this study is to determine the effect different sources and forms of discretionary foods have on stress perception in healthy adults in a free living, real world setting.

Rationale:

The rationale for conducting this study is to test the effects of sugar-sweetened beverages and grain-based desserts have on perceived health and stress perception, since the evidence for this topic is limited.

ELIGIBILITY:
Inclusion Criteria:

* Adults who consume sugar sweetened beverages and grain based desserts and candy on a regular basis
* Free from major illnesses or chronic disease
* Willing to consume amount of beverages and food provided to supplement usual dietary habits during each period

Exclusion Criteria:

* Recently lost a significant amount or looking to lose weight
* Recently begun a new diet or exercise regimen
* Pregnant or nursing women
* Report restrained eater or having less than 51% control over food preparation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Stress Perception | 12 weeks
  A questionnaire adapted from the SF-12 will be used to measure stress perception.

SECONDARY OUTCOMES:
Body Weight | 12 weeks
  A digital scale will be used to measure body weight.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Odegaard, Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota West Bank Office Building, Minneapolis, Minnesota, United States